CLINICAL TRIAL: NCT00921934
Title: PASCORBIN 7.5g in the Treatment of Viral Infection, Especially Varicella Zoster Infection: An Observational Cohort Study
Brief Title: Intravenous Vitamin C in the Treatment of Viral Infection, Especially in the Treatment of Shingles
Acronym: 168
Status: Completed | Type: Observational
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Collaborators: Dr. Loges & Co. GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 168 A 08 VC
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-11

CONDITIONS: Virus Diseases; Herpes Zoster
Keywords: Herpes; Shingles; virus disease; vitamin C; ascorbic acid; antioxidant; oxidative stress
MeSH Terms: conditions — Virus Diseases; Herpes Zoster; Herpes Simplex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vitamin C: Adult patients suffering from acute viral infection, especially herpes zoster, presenting themselves in Primary Care Centers or hospitals all over Germany, and who are treated with standard therapy and add-on vitamin C.

SUMMARY:
Chronic viral infections induce oxidative stress that can cause a number of concomitant diseases, e.g. cardio-vascular diseases or metabolic disorders. Therefore, a sufficient treatment of oxidative stress may be of benefit for the patient to prevent further diseases.

Shingles (herpes zoster infection) have been successfully treated with antioxidative substances like high-dose vitamin C for ages. Not only the acute symptoms can be diminished by high-dose vitamin C. Even long-term sequelae, like painful post-herpetic neuropathy, may be mitigated or even fully avoided.

ELIGIBILITY:
Due to the design of an Observational Cohort Study, no inclusion or exclusion criteria are named. The included patient group is described under "Cohort / Group".

Observational Criteria:

* adult patients
* acute viral infection (especially herpes zoster)
* Primary Care patient
* eligible for add-on therapy with vitamin C
* willingness to provide pseudonymized data to the Sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of adult patients suffering from acute viral infections, especially herpes zoster, presenting themselves in Primary Care Centers or hospitals all over Germany.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schencking, MD, Principal Investigator — Rheinstr. 77a, D-56235 Ransbach-Baumbach; Bianka Krick, Study Director — Pascoe Pharmazeutische Praeparate GmbH
Locations (1):
- Praxis Dr. Schencking, Rheinstr. 77a, Ransbach-Baumbach, Rhineland-Palatinate, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited from general practioners between April 2009 and December 2010.
Pre-assignment Details: Between April 2009 and December 2010 16 general practitioners recorded data of 68 participants with symptomatic herpes zoster (one patient with viral infection) who received vitamin C intravenously (Pascorbin® 7.5 g/50 ml) for approximately 2 weeks in addition to standard treatment.
Period: Overall Study
Arm/Group | Vitamin C
Started | 68
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin C
Number analyzed (Participants) | 68
Age, Customized [Mean (Standard Deviation); unit: years]
  Between 18 and 65 years | 43.6 (14.5)
  >=65 years | 67.7 (8.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — zero patients were analyzed in this age group
  Between 18 and 65 years | 44
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 29
Region of Enrollment [Number; unit: participants]
  Germany | 68
Body mass index [Mean (Standard Deviation); unit: kg/m^2]
  Female | 24.4 (3.9)
  Male | 27.6 (4.9)
  Total | 25.8 (4.6)
Weihgt, kg [Mean (Standard Deviation); unit: kg]
  Female | 65.6 (10.6)
  Male | 83.3 (12.4)
  Total | 73.1 (14.3)
Concomitant immunosuppressive disease [Number; unit: participants] — Immunosuppressive conditions = malignant neoformation of the mammae, diabetes mellitus, bronchial asthma, neurodermatitis, malignant neoformation, chemotherapy, breast ablation, hyperthyreosis, B-cell lymphoma, laryngeal cancer, pernicious anaemia, hepatitis, non-Hodgkin lymphoma, immunoglobulin-G deficiency, pneumoconiosis.
  participants
    yes | 11
    no | 57
Duration of Herpes Zoster-specific complaints (separated into groups) [Number; unit: participants]
  0 to 14 days | 31
  2 to 6 weeks | 30
  > 6 weeks | 7
Number of concomitant medications for the inclusion diagnosis [Number; unit: participants]
  None | 24
  1 | 24
  2 | 15
  3 | 2
  4 | 3
Common symptoms at baseline gerneral fatigue [Number; unit: participants]
  Not present | 13
  Mild | 30
  Moderate | 20
  Strong | 5
Common symptoms at baseline impaired concentration [Number; unit: participants]
  Not present | 24
  Mild | 24
  Moderate | 17
  Strong | 3

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain Measured by VAS
Description: VAS (minimum = 0 = no pain, maximum = 10 = extrem pain, change of pain measured by VAS
Time Frame: visit 1 - 3
Population: Three patients had no pain at baseline (score value = 0) and were thus excluded from the statistical analysis. The descriptive results per visit are presented in the data below. V1 (Baseline) N=64, V2 (week 2)N=64, V3 (week 12)N= 47, Last vsit (N=64).
Measure: Mean (Standard Deviation); unit: pain intensity
Arm/Group | Vitamin C
Number analyzed (Participants) | 68
pain intensity
  V1 (Baseline) | 5.8 (2.4)
  V2 (week 2) | 2.2 (2.2)
  V3 (week 12) | 0.6 (1.1)
  Last visit | 1.2 (2.0)

ADVERSE EVENTS:
Time Frame: 1.5 years
Arm/Group | Vitamin C
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 2/68
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin C (N=68)
Sensation of heat on the injection site (Nervous system disorders) | 1 (1)
numbness sensation up to the fingertips (Nervous system disorders) | 1 (1)
burning (Nervous system disorders) | 1 (1)
Urticarial drug inducted exanthema on truncus (Skin and subcutaneous tissue disorders) | 1 (1)
Urticarial drug inducted exanthema on torso (Skin and subcutaneous tissue disorders) | 1 (1)
protracted diarrhoe (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No